CLINICAL TRIAL: NCT00501072
Title: Use of a Real Time Continuous Glucose Monitoring System (RT-CGMS) in Type 1 Diabetes Patients on Continuous Intraperitoneal Insulin Infusion (CIPII. A Feasibility Study
Brief Title: Safety and Efficacy of RT-CGMS in Patients With Type 1 Diabetes Mellitus Treated With an Implantable Pump
Acronym: IP_RT-CGMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Foundation, The Netherlands (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07.0644; NL12530.075.06
Record Dates: First submitted 2007-07-12; First posted 2007-07-13 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: hyperglycemia; hypoglycemia; glucose variability; insulin infusion system; implantable insulin pump; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open (Experimental): Real-Time Continuous Glucose monitoring System (RT-CGMS) with alarm setting active and ability to view glucose trend profiles
  Interventions: Device: Real-Time Continuous Glucose monitoring System (RT-CGMS)
- Blind (No Intervention): RT-CGMS is applied without alarm setting and without the ability to watch glucose trend profiles

INTERVENTIONS:
Device: Real-Time Continuous Glucose monitoring System (RT-CGMS)
  Arms: Open

SUMMARY:
To investigate the effectiveness and safety of a Real Time Continuous Glucose Monitoring System (RT-CGMS in a population of patients with type 1 diabetes mellitus treated with insulin through an implanted pump.

DETAILED DESCRIPTION:
Background: Strict glycaemic control reduces risk of complications and improves quality of life in patients with type 1 diabetes mellitus. Real Time Continuous Glucose Monitoring System (RT-CGMS) is a novel system which can provide patients and health care professionals with real time information about the blood glucose level without the need for multiple invasive measurements. Furthermore, with continuous monitoring it is possible to identify trends in glycaemic profiles. Its effectiveness and safety have never been tested in a population of patients with type 1 diabetes mellitus treated with insulin through an implanted pump.

Objective: To investigate the effectiveness and safety of the RT-CGMS in patients treated with intraperitoneal continuous insulin infusion (CIPII).

Study design: Open label, randomized cross-over, single-center controlled trial.

Study population: Patients on CIPII. Intervention: There are 3 study phases. In the Baseline phase, all patients will have the RT-CGMS blinded so that no information on blood glucose values measured and stored by the RT-CGMS will be available to care-givers, investigators or patients during this study period. Randomization will determine the sequence of blinded and unblinded RT-CGMS in the 2nd and 3rd phase. When the RT-CGMS is not blinded, the system will alert whenever a glucose level falls below or rises above preset values. Sensor values are not intended to be used directly for making therapy adjustments. Whenever a value is below or above the preset value, the blood glucose level will be measured using a blood glucose meter and therapy adjustments based on this value will be done according to protocol.

Study endpoints: Primary: Percentage of time spent in euglycaemia. Secondary: percentage of time spent in hypoglycaemia and hyperglycaemia, incidence and severity of hypoglycaemia (as measured with SMBG), incidence of adverse effects, number of measurements of blood glucose (SMBG) performed, number of adjustments of insulin therapy, patient satisfaction, agreement of paired SMBG and RT-CGMS measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients on CIPII and treated in the Isala Clinics, Zwolle, The Netherlands
* Age >18 years
* Uncontrolled diabetes mellitus type 1

Exclusion Criteria:

* Failure to obtain informed consent
* Any condition prevention proper handling of the device, for instance hearing impairment or visual impairment
* Known allergy to sensor (parts)
* Currently pregnant or trying to conceive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Clinical effectiveness: percentage of time spent in euglycaemia | 3-6 days

SECONDARY OUTCOMES:
Clinical effectiveness: Percentage of time spent in hypoglycaemia and hyperglycaemia. | 3-6 days
Safety: incidence of adverse effects | ca. 30 days
Incidence of hypoglycaemia; Number of SMBG performed, Number of adjustments of insulin therapy, Patient satisfaction, agreement of paired SMBG and RT-CGMS measurements. | 3-6 -30 days

CONTACTS AND LOCATIONS:
Overall Officials: Henk J Bilo, MD PhD, FRCP, Principal Investigator — Isala Clinics, Diabetes Centre and University Medical Center Groningen
Locations (1):
- Diabetes Outpatient Clinic, Isala clinics, Zwolle, Netherlands

REFERENCES:
- [Derived] Logtenberg SJ, Kleefstra N, Groenier KH, Gans RO, Bilo HJ. Use of short-term real-time continuous glucose monitoring in type 1 diabetes patients on continuous intraperitoneal insulin infusion: a feasibility study. Diabetes Technol Ther. 2009 May;11(5):293-9. doi: 10.1089/dia.2008.0088. PMID 19425877